CLINICAL TRIAL: NCT06058676
Title: A Controlled Clinical Study of Prediction of Cerebral Hyperperfusion Syndrome After Carotid Artery Stenting by Using Multi-parameter Characteristics Based on Cerebral Autoregulation
Brief Title: Prediction of Hyperperfusion After Carotid Stenting by Multi-parameter Characteristics Based on Cerebral Autoregulation
Acronym: HACASS
Status: Enrolling by invitation | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-9-15
Record Dates: First submitted 2023-09-21; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Cerebral Artery Stenosis; Carotid Artery Stent; Dynamic Cerebral Autoregulation
Keywords: Ultrasonography; Carotid artery stent; Dynamic cerebral autoregulation; Cerebral hyperperfusion; Hemodynamics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with reduced cerebrovascular reserve: Interventions:
  Procedure: carotid artery stenting
  Interventions: Procedure: carotid artery stenting
- Patients with sufficient cerebrovascular reserve: Interventions:
  Procedure: carotid artery stenting
  Interventions: Procedure: carotid artery stenting

INTERVENTIONS:
Procedure: carotid artery stenting — The procedures will be performed for patients with general or local anesthesia. Implantation of stents at the site of carotid artery stenosis for the treatment of carotid severe stenosis. A suitable balloon will be selected based on the internal carotid arterial（ICA）diameter, as shown on the digital subtraction angiography（DSA）image. The use of a balloon for predilatation or postdilatation depends on the degree of stenosis. The type of stent will be selected according to several factors, such as the length and configuration of the lesion, vascular morphology, vessel diameter, plaque characteristics, stent characteristics, and surgeon experience.

SUMMARY:
Cerebral hyperperfusion syndrome (CHS) is one of the severe complication after carotid artery stenting with a high mortality rate. CHS was defined as cerebral hyperperfusion (CH) with clinical symptoms such as unilateral headache, convulsions, hemiparesis/hemiplegia, visual disturbances, ataxia, aphasia, while CH could be a disastrous outcome causing complication after carotid revascularization if not managed properly and timely.

This is a single-center prospective cohort study to investigate the risks of CH after carotid artery stenting. All patients with severe carotid artery stenosis underwent carotid arterial ultrasonography and dynamic cerebral autoregulation (dCA) test by transcranial Doppler sonography (TCD) before operation. The postoperative carotid ultrasound and transcranial Doppler sonography (TCD) results are also needed. The investigators will collect this test data at 48h, 1 month and 3months after carotid artery stenting（CAS）. According to the examination results, they were divided into two groups: CH group and non-CH group.

The investigators will collect data before CAS, on all participants' age, sex, heart rate, BP and end-tidal carbon dioxide (ET-CO2) and the following information from the patients : (i)demographic data, such as hypertension, coronary heart disease, diabetes, hyperlipidemia, smoking and body mass index; (ii) relevant clinical symptoms; (iii) preoperative colour Doppler ultrasonography（CDU）and transcranial Doppler sonography(TCD) results; (iv) The cerebral blood flow velocity (CBFV) of the middle cerebral artery（MCA） induced will be measured by non-invasively and continuously dCA test.

This study could be aimed to analyze the factors influencing cerebral hyperperfusion after CAS. The purpose of this study will be to perform more precise risk stratification for high-risk CH patients and improve the quality of life of them.

Statistical Analysis The Statistical Package for the Social Sciences（SPSS）software Version 26.0 (IBM, New York, USA) will be used for statistical analyses. The indicators with P < 0.2 in the univariate analysis will be entered into a logistic regression analysis to investigate the independent risk factors for CH after CAS. All tests will be performed two sided, and a P < 0.05 will be considered statistically significant.

DETAILED DESCRIPTION:
1. To analysis the incidence of postoperative complications such as CH and CHS within 1 months and to find the risk factors of CH.

   A. To enroll 400 cases of patients suffering from carotid artery stenosis. the investigators perform TCD on patients by Sonographer for identifying CH.

   B. Postoperative CH will be defined in patients whose MCA mean velocity increased by more than 100% within 48 hour after carotid artery stent.

   C. CH and CHS mostly occurs within one week after CAS. Although there are a few reports of CHS occurring from three weeks to four weeks after CAS.

   D. All tests are non-invasive.
2. The diagnosis of CHS will be based on the following criteria:

   A. The appearance of symptoms within 1 month after surgery.

   B. First-time unilateral headache, convulsions, hemiparesis/hemiplegia, visual disturbances, ataxia, aphasia, signs of cerebral edema or intracerebral hemorrhage.

   C. Increase in cerebral blood flow in the middle cerebral artery > 100% compared to the preoperative value measured by transcranial dopplerography.

   D. Hypertensive encephalopathy, reversible posterior leukoencephalopathy syndrome and reversible cerebral vasoconstriction syndrome are excluded.
3. The parameter of ultrasonic measurement

A. The CDU before CAS about plaque imaging and other parameters will be stored in Statistical Package for the Social Sciences （PACS）and analyzed later.

B.The TCD peri-CAS will be used to detect main intracranial arteries, the peak systolic velocity（PSV）, end-diastolic velocity（EDV）and PI of bilateral MCA will be recorded.

C.The post-CAS imaging and parameters included the characteristics of stent and hemodynamic parameters by CDU and TCD.

ELIGIBILITY:
Inclusion Criteria:

* (1) Male and non-pregnant, non-breastfeeding female subjects whose age is ≥ 18 years and ≤ 80.

  (2) Symptomatic patients with internal carotid artery stenosis≥50% on angiography, or asymptomatic patients with internal carotid artery stenosis≥70% on angiography treatable with carotid artery stenting.

  (3) Patient is willing and capable of complying with all study protocol requirements, including the specified follow-up visits and can be contacted by telephone.

Exclusion Criteria:

* (1) Patients with severe carotid artery stenosis caused by non-atherosclerosis diseases, such as dissection or arteritis.

  (2) Inability to cooperate with all this examination.

  (3) Patients without complete clinical or imaging information.

  (4) Patients not evaluated by CDU before CAS or within 1 week after CAS.

  (5) Lack of follow up with CDU after CAS.

  (6) Patients with poor temporal sound window or closure of the temporal window.

  (7) Hyperthyroidism, hemicrania, severe arrhythmia and other diseases affecting dCA.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients 18 years of age and older. Symptomatic patients with internal carotid artery stenosis≥50% on angiography, or asymptomatic patients with internal carotid artery stenosis≥70% on angiography.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Cerebral hyperperfusion | within 7 days post-operation
  Postoperative CH will be defined in patients whose MCA mean velocity increased by more than 100% after carotid artery stent.

SECONDARY OUTCOMES:
Cerebral hyperperfusion syndrome | with 1 month post-operation
  CHS always occurs after CAS of high-grade carotid artery stenosis causing cerebral hemodynamic insufficience. CHS was defined as a clinical triad of ipsilateral head ache, seizures, and neurologic deficits in the absence of cerebral ischemia after a successful carotid stenting.
Major stroke | within 7 days post-operation
  The incidence of major stroke after CAS, defined as new onset of neurological symptoms causing an increase of NIHSS ≥ 4 or worsening of existing focal neurological deficit lasting ≥ 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: yingqi Xing, MD, Principal Investigator — Department of Vascular Ultrasonography, Xuanwu Hospital. Beijing Institute of Brain Disorders.
Locations (1):
- Department of Vascular Ultrasonography, Xuanwu Hospital of Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bonow RH, Young CC, Bass DI, Moore A, Levitt MR. Transcranial Doppler ultrasonography in neurological surgery and neurocritical care. Neurosurg Focus. 2019 Dec 1;47(6):E2. doi: 10.3171/2019.9.FOCUS19611. PMID 31786564
- [Background] Liu Y, Tarumi T, Liu B, Li J, Wu X, Zhang N, Hua Y. Dynamic Cerebral Autoregulation in Preclinical Atherosclerotic Cardiovascular Disease. J Stroke Cerebrovasc Dis. 2020 Jun;29(6):104810. doi: 10.1016/j.jstrokecerebrovasdis.2020.104810. Epub 2020 Apr 11. PMID 32291129
- [Background] Panerai RB, Brassard P, Burma JS, Castro P, Claassen JA, van Lieshout JJ, Liu J, Lucas SJ, Minhas JS, Mitsis GD, Nogueira RC, Ogoh S, Payne SJ, Rickards CA, Robertson AD, Rodrigues GD, Smirl JD, Simpson DM; Cerebrovascular Research Network (CARNet). Transfer function analysis of dynamic cerebral autoregulation: A CARNet white paper 2022 update. J Cereb Blood Flow Metab. 2023 Jan;43(1):3-25. doi: 10.1177/0271678X221119760. Epub 2022 Aug 12. PMID 35962478